CLINICAL TRIAL: NCT03248128
Title: A Randomised, Double-blind, Parallel Group, Multicentre, Stratified, Study Evaluating the Efficacy and Safety of Once Daily Fluticasone Furoate/Vilanterol Inhalation Powder Compared to Once Daily Fluticasone Furoate Inhalation Powder in the Treatment of Asthma in Participants Aged 5 to 17 Years Old (Inclusive) Currently Uncontrolled on Inhaled Corticosteroids
Brief Title: Safety and Efficacy Study of Fluticasone Furoate/Vilanterol (FF/VI) Fixed Dose Combination (FDC) Compared to FF Alone in Subjects With Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 107116; 2016-004086-87 (EudraCT Number)
Record Dates: First submitted 2017-08-09; First posted 2017-08-14 (Actual); Results first posted 2022-10-12 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Asthma
Keywords: Fluticasone furoate; Efficacy; Vilanterol; Asthma; Safety; GW642444; GW685698
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to receive FDC of FF/VI inhalation powder compared to FF inhalation powder, once daily in cohort A and cohort B.
Who Masked: Participant, Investigator
Masking Description: This will be a double blind study. Subjects and investigator will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Subjects receiving FF/VI in cohort A (Experimental): Subjects will be randomized in 1:1 ratio to receive a FDC of FF/VI with a dose of 50/25 mcg administered once daily in the morning via ELLIPTA DPI.
  Interventions: Drug: FF/VI via ELLIPTA DPI
- Subjects receiving FF in cohort A (Active Comparator): Subjects will be randomized in 1:1 ratio to receive FF with a dose of 50 mcg administered once daily in the morning via ELLIPTA DPI.
  Interventions: Drug: FF via ELLIPTA DPI
- Subjects receiving FF/VI in cohort B (Experimental): Subjects will be randomized in 1:1 ratio to receive a FDC of FF/VI with a dose of 100/25 mcg administered once daily in the morning via ELLIPTA DPI.
  Interventions: Drug: FF/VI via ELLIPTA DPI
- Subjects receiving FF in cohort B (Active Comparator): Subjects will be randomized in 1:1 ratio to receive FF with a dose of 100 mcg administered once daily in the morning via ELLIPTA DPI.
  Interventions: Drug: FF via ELLIPTA DPI

INTERVENTIONS:
Drug: FF/VI via ELLIPTA DPI — ELLIPTA DPI inhaler will contain two individual blister strips; the first strip will contain FF(50 or 100 mcg) and second strip will contain VI (25 mcg).
  Arms: Subjects receiving FF/VI in cohort A; Subjects receiving FF/VI in cohort B
Drug: FF via ELLIPTA DPI — ELLIPTA DPI inhaler will contain a single blister strip of FF (50 or 100 mcg).
  Arms: Subjects receiving FF in cohort A; Subjects receiving FF in cohort B

SUMMARY:
The goal of asthma treatment is to achieve and maintain asthma control and to reduce the future risk of exacerbations. Inhaled corticosteroids (ICS) are considered as the most effective anti- inflammatory treatment for all severities of persistent asthma. For children >=5 years of age and adolescents whose asthma is uncontrolled, low-dose ICS plus adjunctive therapy with long-acting beta agonist (LABA) is considered as effective. Thus, this study is designed to evaluate the efficacy and safety of FF (ICS component)/VI (LABA component) compared to FF alone for the treatment of asthma, in subjects aged 5 to 17 years old currently uncontrolled on ICS. The study will be conducted over a total duration of approximately 29 weeks: 4 week run-in period, 24-week double-blind treatment period and 1-week follow-up period. Subjects will be randomized to receive FDC of FF/VI or FF administered via ELLIPTA® dry powder inhaler (DPI). The dose of both FF/VI and FF alone will be selected based on the age of subjects. Subjects will receive a short acting beta 2 agonist (SABA) (albuterol /salbutamol) as a rescue medication throughout the study. A total of 870 subjects will be randomized in the study. Of this, 652 subjects will be aged 5 to 11 years (cohort A), and 218 will be aged 12 to 17 years inclusive (cohort B). ELLIPTA is a registered trademark of GlaxoSmithKline (GSK) group of companies.

ELIGIBILITY:
Inclusion Criteria:

* For all subjects: Between 5 and 17 years of age inclusive, at the time of signing the informed consent.
* A history of symptoms consistent with a diagnosis of asthma for at least 6 months.
* Pre-bronchodilator FEV1 >50 percent to <=90 percent predicted normal. A minimum of 2 efforts that are considered acceptable (not necessarily repeatable) are required to be eligible.
* Lung function reversibility defined as an increase of >=12 percent in FEV1 within 10 to 40 minutes following 2 to 4 inhalations of salbutamol inhalation aerosol (or 1 nebulized treatment with albuterol/salbutamol solution). Use of a spacer is permitted.
* Uncontrolled asthma, with a childhood asthma control test (cACT)/ACT score <=19.
* Receiving stable asthma therapy (SABA inhaler plus ICS [total daily dose <=FP 250 micrograms (mcg) or equivalent]) for at least 4 weeks prior to Visit 1 (i.e. screening).
* Able to replace their current SABA treatment with salbutamol aerosol inhaler at Visit 1 for use as needed for the duration of the study. Salbutamol metered dose inhaler (MDI) will be administered with or without a spacer, to be used as determined by the investigator. The use or non-use of the spacer should be consistent for an individual subject throughout the study.
* Male or female subjects will be included. Females of reproductive potential must agree to follow 1 of the options listed (which include abstinence) in the Modified List of Highly Effective Methods for Avoiding Pregnancy in Females of Reproductive Potential (FRP) from 30 days prior to the first dose of study medication and until at least five terminal half-lives or until any continuing pharmacologic effect has ended, whichever is longer after the last dose of study medication and completion of the follow-up call. The investigator is responsible for ensuring that subjects understand how to properly use these methods of contraception.
* Written informed consent from at least 1 parent/care giver (legal guardian) and accompanying informed assent from the subject (where the subject is able to provide assent) prior to admission to the study. If applicable, subject must be able and willing to give assent to take part in the study according to the local requirement. The study investigator is accountable for determining a child's capacity to assent to participation in a research study, taking into consideration any standards set by the responsible independent ethics committee (IEC); subject and their legal guardian(s) understand that the study requires them to be treated on an outpatient basis; subject and their legal guardian(s) understand that they must comply with study medication and study assessments including recording of PEF and rescue SABA use, attending scheduled study visits, and being accessible by a telephone call.
* For subjects eligible for randomization; asthma control: uncontrolled asthma, with a cACT/ACT score <=19.
* A technically acceptable pre-bronchodilator FEV1 >50 percent to <=90 percent predicted normal at Visit 2. A minimum of 2 efforts that are considered acceptable and repeatable following the over read are required to be eligible.
* Symptoms and rescue use: demonstrated and reported in a daily diary symptoms of asthma (a score of >=1 on the day-time or night-time asthma symptom scores) and/or daily albuterol/salbutamol on at least 3 of the last 7 consecutive days of the run-in period (not including the date of randomization).
* Compliance with run-in medication: compliance is defined as use of run-in medication on at least 4 of the last 7 consecutive days of the run-in period (not including the date of randomization) recorded in the electronic subject diary.
* Compliance with completion of the daily diary reporting: defined as completion of all questions on 4 out of the last 7 days during the run-in period (not including the date of randomization).

Exclusion Criteria:

* For all subjects: History of life threatening asthma defined as an asthma episode that required intubation and/or was associated with hypercapnea, respiratory arrest or hypoxic seizures.
* Any asthma exacerbation requiring the use of oral steroids within 6 weeks of Visit 1, systemic or depot corticosteroids within 12 weeks of Visit 1, or ER attendance within 3 months of Visit 1 or hospitalization within 6 months of Visit 1.
* A culture documented or suspected bacterial or viral infection of the upper or lower respiratory tract, sinus or middle ear that has not resolved within 4 weeks of Visit 1 and which led to a change in asthma management or, in the opinion of the investigator, is expected to affect the subject's asthma status or the subject's ability to participate in the study.
* Clinical visual evidence of oropharyngeal candidiasis.
* Fasting blood glucose at screening >100 milligrams/deciliter (mg/dL) (5.6 moles per liter [mol/L]).
* Obesity (Body Mass Index [BMI] above the 97th centile based on the centers for disease control and prevention [CDC] charts).
* Any significant abnormality or medical condition identified at the screening medical assessment (including serious psychological disorder) that in the investigator's opinion, preclude entry into the study due to risk to the subject or that may interfere with the conduct and/or outcome of the study.
* QTc >450 milliseconds (msec) or QTc >480 msec in subjects with bundle branch block or any other clinically significant abnormality in the screening 12-lead ECG.
* Use of any prohibited medications.
* Present use of any tobacco products.
* Drug allergies: any adverse reaction including immediate or delayed hypersensitivity to any beta 2-agonists, sympathomimetic drug or any intranasal, inhaled, or systemic corticosteroid therapy. Known or suspected sensitivity to the constituents of the ELLIPTA Inhaler (i.e. lactose or magnesium stearate).
* Milk Protein Allergy: history of severe milk protein allergy.
* Participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, five half-lives or twice the duration of the biological effect of the study treatment (whichever is longer).
* Exposure to more than 4 investigational medicinal products within 12 months prior to the first dosing day.
* An affiliation with the investigator site: the parents/guardians or child is an immediate family member of the participating investigator, sub-investigator, study coordinator, or employee of the participating investigator.
* The parent or guardian has a history of psychiatric disease, intellectual deficiency, substance abuse or other condition (example, inability to read, comprehend or write) which may affect: validity of consent to participate in the study; adequate supervision of the subject during the study; compliance of subject with study medication and study procedures (example, completion of daily diary, attending scheduled clinic visits); subject safety and well-being.
* Children in care: children who are wards of the government or state are not eligible for participation in this study.
* For subjects eligible for randomization; Changes in asthma medication that occur after screening.
* Occurrence of a culture-documented or suspected bacterial or viral infection of the upper or lower respiratory tract, sinus or middle ear during the run-in period that led to a change in asthma management or, in the opinion of the investigator, is expected to affect the subject's asthma status or the subject's ability to participate in the study.
* Evidence of an exacerbation, defined as a: deterioration of asthma requiring the use of oral corticosteroids for at least 3 days, or a depot corticosteroid injection, or an in-patient hospitalization due to asthma that required systemic corticosteroids between screening and randomization.
* Clinical visual evidence of oropharyngeal candidiasis at the randomization Visit.
* Unable to use the ELLIPTA inhaler correctly.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 906 (Actual)
Dates: Start 2017-10-20 (Actual); Primary Completion 2022-03-21 (Actual); Study Completion 2022-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (139):
- United States (41):
  - GSK Investigational Site, Hoover, Alabama
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Riverside, California
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Aventura, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Miami Lakes, Florida
  - GSK Investigational Site, Ocala, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Gainesville, Georgia
  - GSK Investigational Site, Savannah, Georgia
  - GSK Investigational Site, Evanston, Illinois
  - GSK Investigational Site, Oak Park, Illinois
  - GSK Investigational Site, Evansville, Indiana
  - GSK Investigational Site, Owensboro, Kentucky
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, White Marsh, Maryland
  - GSK Investigational Site, Ypsilanti, Michigan
  - GSK Investigational Site, Piscataway, New Jersey
  - GSK Investigational Site, Verona, New Jersey
  - GSK Investigational Site, Great Neck, New York
  - GSK Investigational Site, New Hartford, New York
  - GSK Investigational Site, Asheville, North Carolina
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Grove City, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Wexford, Pennsylvania
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Orangeburg, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Summerville, South Carolina
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Lewisville, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Waco, Texas
  - GSK Investigational Site, Murray, Utah
- Argentina (13):
  - GSK Investigational Site, Berazategui, Buenos Aires
  - GSK Investigational Site, CABA, Buenos Aires
  - GSK Investigational Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - GSK Investigational Site, Florida, Buenos Aires
  - GSK Investigational Site, La Plata, Buenos Aires
  - GSK Investigational Site, Lanús, Buenos Aires
  - GSK Investigational Site, Lobos, Buenos Aires
  - GSK Investigational Site, Mar del Plata, Buenos Aires
  - GSK Investigational Site, Nueve de Julio, Buenos Aires
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Mendoza
  - GSK Investigational Site, Rosario
  - GSK Investigational Site, Santa Fe
- Bulgaria (3):
  - GSK Investigational Site, Rousse
  - GSK Investigational Site, Sofia
  - GSK Investigational Site, Stara Zagora
- Canada (3):
  - GSK Investigational Site, Brampton, Ontario
  - GSK Investigational Site, Windsor, Ontario
  - GSK Investigational Site, Québec
- China (2):
  - GSK Investigational Site, Panzhihua, Sichuan
  - GSK Investigational Site, Taiyuan
- Germany (4):
  - GSK Investigational Site, Heidelberg, Baden-Wurttemberg
  - GSK Investigational Site, Mannheim, Baden-Wurttemberg
  - GSK Investigational Site, Rosenheim, Bavaria
  - GSK Investigational Site, Geesthacht, Schleswig-Holstein
- Hungary (2):
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Szeged
- Italy (7):
  - GSK Investigational Site, Parma, Emilia-Romagna
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Bergamo, Lombardy
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Palermo, Sicily
  - GSK Investigational Site, Ancona, The Marches
  - GSK Investigational Site, Perugia, Umbria
- Japan (9):
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Fukui
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Hiroshima
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Tokyo
- GSK Investigational Site, Vilnius, Lithuania
- Mexico (4):
  - GSK Investigational Site, Guadalajara, Jalisco
  - GSK Investigational Site, Zapopan, Jalisco
  - GSK Investigational Site, Monterrey, Nuevo León
  - GSK Investigational Site, Villahermosa, Tabasco
- Poland (15):
  - GSK Investigational Site, Bialystok
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Częstochowa
  - GSK Investigational Site, Katowice
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Ostrowiec Świętokrzyski
  - GSK Investigational Site, Ostrów Wielkopolski
  - GSK Investigational Site, Poznan
  - GSK Investigational Site, Skierniewice
  - GSK Investigational Site, Strzelce Opolskie
  - GSK Investigational Site, Tarnów
  - GSK Investigational Site, Warsaw
  - GSK Investigational Site, Wroclaw
  - GSK Investigational Site, Zawadzkie
- Romania (3):
  - GSK Investigational Site, Brasov
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Târgu Mureş
- Russia (15):
  - GSK Investigational Site, Krasnodar
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Omsk
  - GSK Investigational Site, Penza
  - GSK Investigational Site, Perm
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Samara
  - GSK Investigational Site, Saransk
  - GSK Investigational Site, Saratov
  - GSK Investigational Site, St'Petersburg
  - GSK Investigational Site, Tomsk
  - GSK Investigational Site, Ufa
  - GSK Investigational Site, Volgograd
  - GSK Investigational Site, Voronezh
  - GSK Investigational Site, Yaroslavl
- South Africa (14):
  - GSK Investigational Site, Boksburg, Gauteng
  - GSK Investigational Site, Johannesburg, Gauteng
  - GSK Investigational Site, Pretoria, Gauteng
  - GSK Investigational Site, Middelburg, Mpumalanga
  - GSK Investigational Site, Panorama, Western Province
  - GSK Investigational Site, Bellville
  - GSK Investigational Site, Bloemfontein
  - GSK Investigational Site, Cape Town
  - GSK Investigational Site, Durban
  - GSK Investigational Site, eMkhomazi
  - GSK Investigational Site, Pretoria
  - GSK Investigational Site, Somerset West
  - GSK Investigational Site, Soweto
  - GSK Investigational Site, Vosloorus Ext 2
- Spain (3):
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid

IPD SHARING:
Plan to Share IPD: Yes
GSK will assess requests from qualified researchers for anonymized individual patient-level data (IPD) and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD is made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf

REFERENCES:
- [Background] Bareille P, Forth R, Imber V, Bondarenko I, Michaud A, Majorek-Olechowska B. Once-daily fluticasone furoate/vilanterol vs once-daily fluticasone furoate in patients with asthma aged 5 to 17 years. Ann Allergy Asthma Immunol. 2024 Nov;133(5):537-544.e4. doi: 10.1016/j.anai.2024.06.024. Epub 2024 Jun 25. PMID 38936466

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 2402 participants screened, 906 participants were randomized, of which 4 participants did not receive study treatment. 902 participants received at least 1 dose of study medication creating the Intent to treat (ITT) Population.
Groups:
- Participants Who Received Fluticasone Furoate/Vilanterol (FF/ VI) Fixed Dose Combination (FDC): 5-11 years old pediatric population were administered FF/VI as a FDC of 50/25 micrograms (mcg) and the 12-17 years old adolescent population received 100/25 mcg once daily via ELLIPTA dry powder inhaler (DPI). Each participant, in addition used albuterol/salbutamol (inhalation aerosol or nebuliser) as required throughout the entire study period as rescue medication for symptomatic relief of asthma symptoms.
- Participants Who Received FF: 5-11 years old pediatric population were administered FF as a monotherapy of 50 mcg and the 12-17 years old adolescent population received 100 mcg once daily via ELLIPTA DPI. Each participant, in addition used albuterol/salbutamol (inhalation aerosol or nebuliser) as required throughout the entire study period as rescue medication for symptomatic relief of asthma symptoms.
Period: Overall Study
Arm/Group | Participants Who Received Fluticasone Furoate/Vilanterol (FF/ VI) Fixed Dose Combination (FDC) | Participants Who Received FF
Started | 455 | 451
ITT Population | 454 | 448
Completed | 433 | 431
Not Completed | 22 | 20
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 16 | 14
Not completed — Site Closed | 4 | 3
Not completed — Randomized, but did not receive treatment | 1 | 3

BASELINE CHARACTERISTICS:
Population: Baseline Characteristic data are reported for 902 participants who received at least 1 dose of study medication creating the ITT Population.
Groups:
- Participants Who Received FF/ VI FDC: 5-11 years old pediatric population were administered FF/VI as a FDC of 50/25 mcg and the 12-17 years old adolescent population received 100/25 mcg once daily via ELLIPTA DPI. Each participant, in addition used albuterol/salbutamol (inhalation aerosol or nebuliser) as required throughout the entire study period as rescue medication for symptomatic relief of asthma symptoms.
- Total: Total of all reporting groups
Arm/Group | Participants Who Received FF/ VI FDC | Participants Who Received FF | Total
Number analyzed (Participants) | 454 | 448 | 902
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 9.9 (3.02) | 10.0 (2.97) | 10.0 (2.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 165 | 191 | 356
  Male | 289 | 257 | 546
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American/African Heritage | 34 | 40 | 74
  American Indian or Alaska Native | 22 | 29 | 51
  Asian | 32 | 26 | 58
  Multiple | 31 | 33 | 64
  White | 335 | 320 | 655

OUTCOME MEASURES:

1. Primary Outcome: Absolute Weighted Mean of Forced Expiratory Volume in 1 Second (FEV1) (0-4 Hours) at Week 12 in 5-17 Year Old Population
Description: Pulmonary function was measured by FEV1, defined as the maximal amount of air that can be forcefully exhaled in one second using a standardized calibrated spirometer. Weighted mean FEV1 was derived using the post-dose assessments (after 30 minutes and 1, 2, 3, 4 hours) with their actual times and using the pre-dose assessment as the 0 hour measurement.
Time Frame: Week 12
Population: ITT population (5-17 years old) included all randomized participants who received at least one dose of study treatment. Only those participants with data available at the specified time point have been analyzed.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Participants Who Received FF/ VI FDC | Participants Who Received FF
Number analyzed (Participants) | 397 | 399
Liters | 2.082 (0.7598) | 1.994 (0.6998)
Statistical Analysis 1: Comparison: Participants Who Received FF/ VI FDC vs Participants Who Received FF; Test type: Superiority; p < 0.001, ANCOVA; Analysis was performed using ANCOVA with covariates of baseline, region, sex, age and treatment; Least Square Mean Difference = 0.083, 95% CI 2-sided [0.037 to 0.129]

2. Primary Outcome: Change From Baseline in Mean Pre-dose Morning Peak Expiratory Flow (AM PEF) in 5-11 Year Old Population
Description: PEF was defined as the maximum speed of expiration of a participant. PEF was measured using a hand-held electronic peak flow meter each morning prior to the dose of study medication and any rescue albuterol/salbutamol inhalation aerosol use. The best of three measurements were recorded in the electronic patient diary. The mean morning PEF was calculated for each participant as an averaged mean over weeks 1-12 of the treatment period. Baseline was defined as the average of measurements with a non-missing value from Day -6 to Day 1 of pre-dose.
Time Frame: Baseline and Week 1-12
Population: ITT population (5-11 years old) was a subset of the ITT (5-17 years old) population for participants 11 years old and younger at screening (Visit 1). Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Liters per minute (L/min)
Groups:
- Participants Who Received FF/ VI FDC (5-11 Year Old Population): Participants aged 5 to 11 years received FDC of 50 mcg/ 25 mcg dose of FF/VI once daily in the morning via ELLIPTA DPI. Each participant, in addition used albuterol/salbutamol (inhalation aerosol or nebuliser) as required throughout the entire study period as rescue medication for symptomatic relief of asthma symptoms.
- Participants Who Received FF (5-11 Year Old Population): Participants aged 5 to 11 years received 50 mcg dose of FF once daily in the morning via ELLIPTA DPI. Each participant, in addition used albuterol/salbutamol (inhalation aerosol or nebuliser) as required throughout the entire study period as rescue medication for symptomatic relief of asthma symptoms.
Arm/Group | Participants Who Received FF/ VI FDC (5-11 Year Old Population) | Participants Who Received FF (5-11 Year Old Population)
Number analyzed (Participants) | 336 | 335
Liters per minute (L/min) | 11.9 (37.63) | 8.9 (35.62)
Statistical Analysis 1: Comparison: Participants Who Received FF/ VI FDC (5-11 Year Old Population) vs Participants Who Received FF (5-11 Year Old Population); Test type: Superiority; p = 0.228, ANCOVA; Analysis was performed using analysis of covariance (ANCOVA) with covariates of baseline, region, sex, age and treatment; Least Square Mean Difference = 3.2, 95% CI 2-sided [-2.0 to 8.4]

3. Secondary Outcome: Change From Baseline in Mean Pre-dose AM PEF Period in 5-17 Year Old Population
Description: PEF was defined as the maximum speed of expiration of a participant. PEF was measured using a hand-held electronic peak flow meter each morning prior to the dose of study medication and any rescue albuterol/salbutamol inhalation aerosol use. The best of three measurements were recorded in the daily diary. The mean morning PEF was calculated for each participant as an averaged mean over weeks 1-12 of the treatment period. Baseline was defined as the average of measurements with a non-missing value from Day -6 to Day 1 of pre-dose.
Time Frame: Baseline and Week 1-12
Population: ITT population (5-17 years old). Only those participants with data available at specified time points has been analyzed.
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Participants Who Received FF/ VI FDC | Participants Who Received FF
Number analyzed (Participants) | 453 | 447
L/min | 14.9 (39.94) | 9.3 (38.95)
Statistical Analysis 1: Comparison: Participants Who Received FF/ VI FDC vs Participants Who Received FF; Test type: Superiority; p = 0.011, ANCOVA; Analysis was performed using ANCOVA with covariates of baseline, region, sex, age and treatment; Least Square Mean Difference = 6.2, 95% CI 2-sided [1.4 to 10.9]

4. Secondary Outcome: Absolute Weighted Mean of FEV1 (0-4 Hours) at Week 12 in 5-11 Year Old Population
Description: as for outcome 1
Time Frame: Week 12
Population: ITT population (5-11 years old). Only those participants with data available at specified time point have been analyzed.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Participants Who Received FF/ VI FDC (5-11 Year Old Population) | Participants Who Received FF (5-11 Year Old Population)
Number analyzed (Participants) | 289 | 291
Liters | 1.762 (0.4977) | 1.711 (0.4817)
Statistical Analysis 1: Comparison: Participants Who Received FF/ VI FDC (5-11 Year Old Population) vs Participants Who Received FF (5-11 Year Old Population); Test type: Superiority; p = 0.002, ANCOVA; Analysis was performed using ANCOVA with covariates of baseline, region, sex, age and treatment; Least Square Mean Difference = 0.073, 95% CI 2-sided [0.028 to 0.118]

5. Secondary Outcome: Change From Baseline in the Percentage of Rescue-free 24-hour Periods Over Weeks 1-12 of the Treatment Period in 5-17 Year Old Population
Description: The number of inhalations of rescue albuterol/salbutamol aerosol used during the day and night were recorded in a daily electronic diary. Percentages of rescue-free 24-hour periods was calculated based on the number of 24-hour periods on which a participant recorded no use of albuterol/salbutamol divided by the length of the time period being assessed (with non-missing values of rescue medication recorded, respectively). A 24-hour period in which the response of participants to both the morning and evening assessments indicated no use of rescue medication was considered as rescue free. Baseline was calculated from the evening (Day -7 to Day -1) and morning (Day -6 to Day 1) measurements. Change from Baseline was calculated as the averaged value during the 12-week treatment period minus the Baseline value.
Time Frame: Baseline and Week 1-12
Population: ITT population (5-17 years old). Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Participants Who Received FF/ VI FDC | Participants Who Received FF
Number analyzed (Participants) | 453 | 447
Percentage | 25.9 (33.78) | 25.8 (36.55)
Statistical Analysis 1: Comparison: Participants Who Received FF/ VI FDC vs Participants Who Received FF; Test type: Superiority; p = 0.870, ANCOVA; Analysis was performed using ANCOVA with covariates of baseline, region, sex, age and treatment; Least Square Mean Difference = -0.3, 95% CI 2-sided [-4.5 to 3.8]

6. Secondary Outcome: Change From Baseline in the Percentage of Symptom-free 24-hour Periods Over Weeks 1-12 of the Treatment Period in 5-17 Year Old Population
Description: The symptom-free days were recorded in a daily electronic diary every day in the morning and evening before taking any rescue or study medication and before the PEF measurement. Percentages of symptom-free 24-hour periods was calculated based on the number of 24-hour periods on which a participant recorded no symptoms divided by the length of the time period being assessed (with non-missing values of rescue medication recorded, respectively). A 24-hour period in which the response of participants to both the morning and evening assessments indicated no symptoms was considered as symptom free. Baseline was calculated from evening (Day -7 to Day -1) and morning (Day -6 to Day 1) measurements. Change from Baseline was calculated as the averaged value during the 12-week treatment period minus the Baseline value.
Time Frame: Baseline and Week 1-12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Participants Who Received FF/ VI FDC | Participants Who Received FF
Number analyzed (Participants) | 453 | 447
Percentage | 25.7 (32.77) | 24.6 (34.62)
Statistical Analysis 1: Comparison: Participants Who Received FF/ VI FDC vs Participants Who Received FF; Test type: Superiority; p = 0.988, ANCOVA; Analysis was performed using ANCOVA with covariates of baseline, region, sex, age and treatment; Least Square Mean Difference = 0.0, 95% CI 2-sided [-4.2 to 4.1]

7. Secondary Outcome: Change From Baseline in Morning (AM) FEV1 at Week 12 in 5-17 Year Old Population
Description: Pulmonary function was measured by FEV1, defined as the maximal amount of air that can be forcefully exhaled in one second. Morning FEV1 was measured using the pre-dose serial spirometry assessment at the Week 12. Baseline was defined as the pre-dose assessment with a non missing value on Visit 2 (Day -5).
Time Frame: Baseline and Week 12
Population: ITT population (5-17 years old). Only those participants with data available at the specified time point has been analyzed.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Participants Who Received FF/ VI FDC | Participants Who Received FF
Number analyzed (Participants) | 417 | 413
Liters | 0.312 (0.3865) | 0.275 (0.3512)
Statistical Analysis 1: Comparison: Participants Who Received FF/ VI FDC vs Participants Who Received FF; Analysis was performed using a repeated measures analysis adjusted for baseline, region, sex, age, treatment, visit, visit by baseline interaction and visit by treatment group interaction; Test type: Superiority; p = 0.124, Repeated measures analysis; Least Square Mean Difference = 0.035, .95% CI 2-sided [-0.010 to 0.080]

8. Secondary Outcome: Change From Baseline in Asthma Control Questionnaire (ACQ-5) Score at Week 24 in 5-17 Year Old Population
Description: Asthma control as measured by improvements in ACQ-5, a five-item questionnaire with response options for each question rated from 0 to 6 scale. A score of 0 indicates well controlled asthma and a score of 6 indicates extremely poorly controlled asthma. Individual questions (concerning nocturnal awakening, waking in the morning, activity limitation, shortness of breath and wheeze) are equally weighted and the ACQ-5 score is calculated as the mean of these 5 item responses. A lower mean score indicates greater asthma control and higher mean score indicates lesser asthma control. Baseline was defined as the pre-dose assessment with a non-missing value on Visit 3 (Day 1).
Time Frame: Baseline and Week 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Participants Who Received FF/ VI FDC | Participants Who Received FF
Number analyzed (Participants) | 385 | 378
Scores on a scale | -1.21 (0.935) | -1.09 (0.976)
Statistical Analysis 1: Comparison: Participants Who Received FF/ VI FDC vs Participants Who Received FF; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.910, Repeated measures analysis; Least Square Mean Difference = -0.01, 95% CI 2-sided [-0.10 to 0.09]

9. Secondary Outcome: Change From Baseline in the Percentage of Rescue-free 24-hour Periods Over Weeks 1-12 of the Treatment Period in 5-11 Year Old Population
Description: as for outcome 5
Time Frame: Baseline and Week 1-12
Population: ITT population (5-11 years old). Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Participants Who Received FF/ VI FDC (5-11 Year Old Population) | Participants Who Received FF (5-11 Year Old Population)
Number analyzed (Participants) | 336 | 335
Percentage | 27.3 (34.4) | 25.6 (37.03)
Statistical Analysis 1: Comparison: Participants Who Received FF/ VI FDC (5-11 Year Old Population) vs Participants Who Received FF (5-11 Year Old Population); Test type: Superiority; p = 0.614, ANCOVA; Analysis performed using ANCOVA with covariates of baseline, region, sex, age and treatment; Least Square Mean Difference = 1.3, 95% CI 2-sided [-3.6 to 6.2]

10. Secondary Outcome: Change From Baseline in the Percentage of Symptom-free 24-hour Periods Over Weeks 1-12 of the Treatment Period in 5-11 Year Old Population
Description: as for outcome 6
Time Frame: Baseline and Week 1-12
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Participants Who Received FF/ VI FDC (5-11 Year Old Population) | Participants Who Received FF (5-11 Year Old Population)
Number analyzed (Participants) | 336 | 335
Percentage | 27.2 (33.16) | 25.8 (34.94)
Statistical Analysis 1: Comparison: Participants Who Received FF/ VI FDC (5-11 Year Old Population) vs Participants Who Received FF (5-11 Year Old Population); Test type: Superiority; p = 0.594, ANCOVA; Analysis was performed using ANCOVA with covariates of baseline, region, sex, age and treatment; Least Square Mean Difference = 1.3, 95% CI 2-sided [-3.6 to 6.3]

11. Secondary Outcome: Change From Baseline in Morning (AM) FEV1 at Week 12 in 5-11 Year Old Population
Description: Pulmonary function was measured by FEV1, defined as the maximal amount of air that can be forcefully exhaled in one second. Morning FEV1 was measured using the pre-dose serial spirometry assessment at the Week 12. Baseline was defined as the pre-dose assessment with a non-missing value on Visit 2 (Day -5).
Time Frame: Baseline and Week 12
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Liters
Groups:
- Participants Who Received FF/ VI FDC (5-11 Year Old Population): Participants aged 5 to 11 years received FDC of 50 mcg/ 25 mcg dose of FF/ VI once daily in the morning via ELLIPTA DPI. Each participant, in addition used albuterol/salbutamol (inhalation aerosol or nebuliser) as required throughout the entire study period as rescue medication for symptomatic relief of asthma symptoms.
Arm/Group | Participants Who Received FF/ VI FDC (5-11 Year Old Population) | Participants Who Received FF (5-11 Year Old Population)
Number analyzed (Participants) | 307 | 304
Liters | 0.263 (0.3029) | 0.245 (0.3192)
Statistical Analysis 1: Comparison: Participants Who Received FF/ VI FDC (5-11 Year Old Population) vs Participants Who Received FF (5-11 Year Old Population); [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.226, Repeated measures analysis; Least Square Mean Difference = 0.028, 95% CI 2-sided [-0.017 to 0.073]

12. Secondary Outcome: Change From Baseline ACQ-5 Score at Week 24 in 5-11 Year Old Population
Description: as for outcome 8
Time Frame: Baseline and Week 24
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Participants Who Received FF/ VI FDC (5-11 Year Old Population) | Participants Who Received FF (5-11 Year Old Population)
Number analyzed (Participants) | 291 | 286
Scores on a scale | -1.25 (0.944) | -1.13 (0.975)
Statistical Analysis 1: Comparison: Participants Who Received FF/ VI FDC (5-11 Year Old Population); [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.663, Repeated measures analysis; Least Square Mean Difference = -0.02, 95% CI 2-sided [-0.13 to 0.09]

13. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) in 5-17 Year Old Population
Description: An AE is any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. SAE is defined as any untoward medical occurrence that, at any dose: results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent disability/incapacity; is a congenital anomaly/birth defect and important medical events may jeopardize the participant or may require medical or surgical intervention/SOC to prevent one of the other outcomes mentioned before.
Time Frame: Up to week 25
Population: ITT (5-17 years old) population
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Who Received FF/ VI FDC | Participants Who Received FF
Number analyzed (Participants) | 454 | 448
Participants
  AEs | 183 | 164
  SAEs | 5 | 5

14. Secondary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Findings in 5-17 Year Old Population
Description: A single 12-lead ECG was obtained using an ECG machine that automatically calculates the heartrate and measures PR, QRS, QT, and QT interval corrected (QTc).
Time Frame: Week 24
Population: ITT population (5-17 years old). Only those participants with data available at the specified time point have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Who Received FF/ VI FDC | Participants Who Received FF
Number analyzed (Participants) | 402 | 398
Participants | 64 | 49

15. Secondary Outcome: Change From Baseline in Fasting Glucose in 5-17 Year Old Population
Description: Blood samples were collected for evaluation of fasting blood glucose pre and post-treatment. Baseline was defined as Visit 1 (Screening).
Time Frame: Baseline and Week 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Participants Who Received FF/ VI FDC | Participants Who Received FF
Number analyzed (Participants) | 370 | 388
mmol/L | -0.12 (0.587) | -0.15 (0.626)

16. Secondary Outcome: Number of Participants With Any Incidence of Asthma Exacerbation Over the 24-week Treatment Period in 5-17 Year Old Population
Description: Asthma exacerbation was defined as deterioration of asthma requiring the use of systemic corticosteroids (tablets, suspension or injection) for at least three days or a single depot corticosteroid injection or an in-patient hospitalization or emergency department visit due to asthma that required systemic corticosteroids.
Time Frame: Up to week 24
Population: ITT population (5-17 years old)
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Who Received FF/ VI FDC | Participants Who Received FF
Number analyzed (Participants) | 454 | 448
Participants | 33 | 38

17. Secondary Outcome: Number of Participants With AEs and SAEs in 5-11 Year Old Population
Description: An AE is any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. SAE is defined as any untoward medical occurrence that, at any dose: results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent disability/incapacity; is a congenital anomaly/birth defect and important medical events may jeopardize the participant or may require medical or surgical intervention/Standard of care (SOC) to prevent one of the other outcomes mentioned before.
Time Frame: Up to week 25
Population: Data only for the ITT (5-11 years old) population have been presented.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Who Received FF/ VI FDC (5-11 Year Old Population) | Participants Who Received FF (5-11 Year Old Population)
Number analyzed (Participants) | 337 | 336
Participants
  AEs | 133 | 122
  SAEs | 4 | 4

18. Secondary Outcome: Number of Participants With Abnormal ECG Findings in 5-11 Year Old Population
Description: A single 12-lead ECG was obtained using an ECG machine that automatically calculates the heartrate and measures PR, QRS, QT, and QTc.
Time Frame: Week 24
Population: ITT population (5-11 years old). Only those participants with data available at the specified time point have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Who Received FF/ VI FDC (5-11 Year Old Population) | Participants Who Received FF (5-11 Year Old Population)
Number analyzed (Participants) | 303 | 298
Participants | 53 | 40

19. Secondary Outcome: Change From Baseline in Fasting Glucose in 5-11 Year Old Population
Description: as for outcome 15
Time Frame: Baseline and Week 24
Population: ITT population (5-11 years old). Only those participants with data available at specified time point have been analyzed.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Participants Who Received FF/ VI FDC (5-11 Year Old Population) | Participants Who Received FF (5-11 Year Old Population)
Number analyzed (Participants) | 274 | 288
mmol/L | -0.13 (0.563) | -0.17 (0.638)

20. Secondary Outcome: Number of Participants With Any Incidence of Asthma Exacerbation Over the 24-week Treatment Period in 5-11 Year Old Population
Description: as for outcome 16
Time Frame: Up to week 24
Population: Data only for the ITT (5-11 years old) population have been presented.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Who Received FF/ VI FDC (5-11 Year Old Population) | Participants Who Received FF (5-11 Year Old Population)
Number analyzed (Participants) | 337 | 336
Participants | 27 | 32

ADVERSE EVENTS:
Time Frame: All cause mortality, Non-serious adverse events (Non-SAEs) and serious adverse events (SAEs) were collected up to 25 weeks (which included one week of follow up contact after completion of the treatment period).
Arm/Group | Participants Who Received FF/ VI FDC | Participants Who Received FF
All-Cause Mortality (participants affected / at risk) | 0/454 | 0/448
Serious Adverse Events (participants affected / at risk) | 5/454 | 5/448
Other Adverse Events (participants affected / at risk) | 107/454 | 71/448
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants Who Received FF/ VI FDC (N=454) | Participants Who Received FF (N=448)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis rotavirus (Infections and infestations) | 1 (1) | 0 (0)
Helicobacter gastritis (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants Who Received FF/ VI FDC (N=454) | Participants Who Received FF (N=448)
Nasopharyngitis (Infections and infestations) | 47 (60) | 34 (42)
Rhinitis (Infections and infestations) | 15 (16) | 6 (6)
Upper respiratory tract infection (Infections and infestations) | 32 (42) | 25 (27)
Headache (Nervous system disorders) | 14 (23) | 9 (13)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 19 (22) | 6 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-08-24): https://cdn.clinicaltrials.gov/large-docs/28/NCT03248128/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-26): https://cdn.clinicaltrials.gov/large-docs/28/NCT03248128/SAP_001.pdf